CLINICAL TRIAL: NCT01415115
Title: A Cross-Sectional Study to Test the Feasibility of Using SCOUT Noninvasive AGE Measurements to Forecast Diabetes Complications
Brief Title: Using SCOUT Noninvasive AGE Measurements to Forecast Diabetes Complications
Acronym: MARC
Status: Completed | Type: Observational
Sponsor: VeraLight, Inc. (Industry)
Collaborators: Medstar Health Research Institute (Other)
Responsible Party: Robert Ratner MD, Medstar Health Research Institute
Other Study IDs: VL-2702
Record Dates: First submitted 2011-08-09; First posted 2011-08-11 (Estimated); Last update posted 2011-08-11 (Estimated); Status verified 2011-08

CONDITIONS: Type 1 Diabetes; Type 2 Diabetes
Keywords: diabetes; hypertension
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Diabetes Mellitus; Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — Blood samples will be drawn for laboratory-based quantification of HbA1c and lipids. Urine samples will be collected to determine urine creatinine and microalbumin
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Type 1 Diabetes: Must have been diagnosed with type 1 diabetes. Subject group will be measured on SCOUT and compared to Type 2 diabetes cohort.
- Type 2 Diabetes: Must have been diagnosed with Type 2 diabetes. This group will be compared to the Type 1 cohort.

SUMMARY:
The trial is designed as a feasibility study to determine the correlation of noninvasive measurements of AGE with the SCOUT device to diabetes complications.

DETAILED DESCRIPTION:
Diabetes mellitus is a major health problem in the United States and throughout the world's developed and developing nations. In 2002, the American Diabetes Association (ADA) has estimated that 12.1 million Americans (4.2%) had been diagnosed with some form of diabetes [1], and the World Health Organization (WHO) assessed the global diabetes caseload at 173 million in the year 2000 [2]. While type 1 patients comprise approximately 5 -10% of the US cases [3], the severe morbidity in those patients including renal failure, blindness, neuropathy and micro- and macro-vascular disease motivate the search for improved techniques for monitoring disease status.

Diabetes is devastating to individual health and has a significant impact on the national economy. In 2002, US economic impact related to diabetes exceeded $132 billion. Due to the numerous complications that result from chronic hyperglycemia a wide array of health services are involved. For example, between 5 and 20 percent of all US services in the areas of cardiovascular disease, kidney disease, endocrine and metabolic complications, and ophthalmic disorders are attributable to diabetes.

Landmark clinical trials in the US and UK have established that tight glucose control via a regimen of glucose monitoring, insulin and/or sulfonylurea or other drug therapy, exercise, and proper diet significantly reduces the progression of, and risk for, developing diabetic complications [4, 5]. Long-term, chronic hyperglycemia is recognized as the initiator of debilitating diabetes-related complications such as blindness, kidney failure and nerve damage [6]. Hence, an effective monitor for overall glycemic control should reflect the long-term, integrated glycemic insult to the body.

One concept of a monitor for long-term glycemic control involves the measurement of an analyte whose concentration monotonically increases over the course of disease progression. Such a chemical marker would not vary with the state in which the patient presented on the day of the test. The process of protein glycation (or 'browning'), governed by the Maillard reaction, produces several advanced glycation endproducts that are attractive candidates for such a 'diabetes meter.' These compounds are currently assayed by invasive procedures, requiring a biopsy specimen, but, based upon initial results with the VeraLight SCOUT, they are also accessible by noninvasive monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Potential subjects for the study will have type 1 or type 2 diabetes. Patients presenting for their periodic examinations at his practice will be given the opportunity to participate. Enrollment will conclude when the target of 250 subjects have been examined.

Exclusion Criteria:

* Wounds or injuries on the volar forearm in the field of view of SCOUT including blisters, cuts, scabs, cracked skin, tattoos and bleeding or oozing skin
* Rash on forearm in field of SCOUT scan including eczema, psoriasis, shingles, rosacea, swimmer's itch, Christmas tree rash, lichen planus, contact dermatitus, ringworm, heat rash or drug rash
* Receiving other investigational treatments
* Receiving medications that may alter skin fluorescence/photosensitivity, including Doxorubicin, Daunomycin, Camptothecin, Protoporphyrin, Fluoroquinolones, Tetracycline and/or Quinidine
* Known to be pregnant
* Prisoner, mentally incompetent or unable to follow study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Potential subjects for the study will have type 1 or type 2 diabetes.
Sampling Method: Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2007-03; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
SCOUT Comparison | 1 day
  This cross-sectional study will test the hypothesis that the correlation between quantitative measurements of skin AGEs by SCOUT noninvasive fluorescence technique, and aggregate diabetic complications, is statistically equivalent to the correlation between the aggregate complications and either disease duration, concurrent HbA1c or individual complications (retinopathy, nephropathy, neuropathy, hypertension and dyslipidemia).

SECONDARY OUTCOMES:
Hypertension | 1 Day
  Five categories of complications--hypertension, dyslipidemia, renal function, retinopathy and neuropathy--will be quantified. Hypertension will be staged based upon blood pressure measurements. The hypertension quantification will follow the classification scheme published by Joint National Committee on Prevention Detection, Evaluation, and Treatment of High Blood Pressure. Dyslipidemia will be quantified by mean plasma lipid values.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Ratner, MD, Principal Investigator — MedStar Health
Locations (1):
- Medstar Health Research Institute, Hyattsville, Maryland, United States